CLINICAL TRIAL: NCT07190339
Title: A Study on the Effectiveness of Pulsed Radiofrequency Treatment Applied to the Femoral and Obturator Nerve Articular Branches Under Ultrasound Guidance in Chronic Hip Osteoarthritis
Brief Title: Femoral and Obturator Nerve Articular Branches Prf
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Supervisor Investigator, Diskapi Teaching and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hip pericapsular nerve pRF
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hip Ostearthritis
Keywords: Pulsed Radiofrequency Treatment; Ultrasonography; femoral and obturator nerve articular branches

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pulsed radiofrequency group (Other): femoral and obturator nerve articular branches pulsed radiofrequency for hip osteoartritis
  Interventions: Procedure: ultrasound-guided femoral and obturator nerve articular branches pulsed radiofrequency

INTERVENTIONS:
Procedure: ultrasound-guided femoral and obturator nerve articular branches pulsed radiofrequency — Hemodynamic monitoring is provided. The hip joint where the procedure will be performed is cleaned with povidone-iodine. Sterile draping is performed. For PRF application to the articular branches of the femoral nerve, a convex ultrasound probe is first used to locate the articular branches of the femoral nerve in the groin area, followed by the articular branches of the obturator nerve. The radiofrequency cannula is inserted sequentially into the target points and sensory feedback is obtained. Then, a pulsed radiofrequency current, which has therapeutic properties for chronic pain and does not damage tissues by exceeding a temperature of 42 degrees, is applied to the relevant nerve root for 240 seconds. Subsequently, an injectate consisting of 2 cc of 5% bupivacaine, 4 mg of dexamethasone, and 2 cc of physiological saline is administered to the same nerve.
  Translated with DeepL.com (free version)

SUMMARY:
In our clinic, patients undergoing pulsed radiofrequency treatment of the femoral and obturator nerve articular branches under ultrasound guidance for pain management due to hip and groin pain associated with hip osteoarthritis will have the efficacy of these methods on pain compared with the Numeric Rating Scale (NRS) and Oxford Hip Score (OHS) at 2, 6, 12 weeks.

DETAILED DESCRIPTION:
Osteoarthritis of the hip joint is a common cause of pain and disability. Patients who do not respond to conservative treatments such as painkillers, physical therapy, and exercise often cannot undergo joint replacement due to comorbid conditions, while some patients prefer to postpone surgery as long as possible. Pulsed radiofrequency treatment applied to the articular branches of the femoral and obturator nerves, which innervate the joint, is a new technique for reducing hip joint pain. Previous studies have reported positive results after applying thermal neurolytic radiofrequency to the target nerves; however, this approach carries the risk of neuritis and neuroma formation. In our study, we aimed to investigate the effectiveness of pRF treatment applied to the articular branches of the femoral and obturator nerves under ultrasound guidance on pain and functionality in patients with chronic hip pain associated with osteoarthritis. The fact that the procedure is performed under ultrasound guidance, does not involve radiation exposure, and is an accessible and easy-to-perform technique makes it preferable for both patients and physicians.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with hip and groin pain who have been diagnosed with hip osteoarthritis by direct radiography
* 2. Patients who have had hip pain above VAS 5 for more than 6 weeks
* 3. Failure of pain treatment with conservative methods such as analgesics and physical therapy

Exclusion Criteria:

* 1. Patients with lumbar radiculopathy and axial back pain, sacroiliac joint, connective tissue disease
* 2. Patients who do not attend follow-up appointments regularly or cannot be reached by phone
* 3. Patients who started additional analgesic medication or underwent additional interventional procedures after the initial interventional procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
numeric rating scale | Change from baseline to 2nd 6 th and 12th weeks after treatment
  The numeric rating scale (NRS) is a pain screening tool, commonly used to assess pain severity at that moment in time using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable"

SECONDARY OUTCOMES:
oxford hip score | Change from baseline to 2nd 6th and 12th weeks after treatment
  The Oxford Hip Score (OHS) is a joint-specific, patient-reported outcome measure designed to assess disability in patients witth hip osteoarthritis

CONTACTS AND LOCATIONS:
Overall Officials: Gevher Rabia Genc Perdecioğlu, Study Chair — Diskapi TRH
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)